CLINICAL TRIAL: NCT05630625
Title: Dynamic Personalized Feedback for Young Adults With a History of Blackout
Brief Title: The Drinking Dashboard Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Mary E Miller, Clinical Psychologist, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2067803
Record Dates: First submitted 2022-11-07; First posted 2022-11-29 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive the Drinking Dashboard or assessment only.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drinking Dashboard (Experimental): Day-level feedback on alcohol use and consequences
  Interventions: Behavioral: Drinking Dashboard
- Assessment Only (No Intervention): Daily assessment control group

INTERVENTIONS:
Behavioral: Drinking Dashboard — Day-level feedback on alcohol use and consequences
  Arms: Drinking Dashboard

SUMMARY:
This study aims to develop and pilot test the efficacy of a "Drinking Dashboard" providing participants weekly feedback on the risk factors and consequences of blackout.

DETAILED DESCRIPTION:
Approximately 50% of young adults who drink alcohol experience alcohol-induced "blackouts," defined as permanent (en bloc) or temporary (fragmentary) memory loss for events that occurred while they are drinking. This experience of alcohol-induced blackout is associated prospectively with alcohol-related harm, including emergency room visits and sexual coercion, with medical care costs exceeding $469,000 per year. While young adults who have recently experienced a blackout report less favorable evaluations of drinking events and increased motivation to decrease their drinking, they do not actually change their drinking behavior as a result of the blackout alone. Collectively, these data suggest that blackouts may serve as an opportunity for intervention, after which young adults are more likely to respond to alcohol feedback. This R34 aims to develop an intervention tailored to individuals who experience blackouts. In the trial phase, 162 young adults (50% female, ≥50% non-college) who report a history of blackout will be randomly assigned to receive the intervention (n=81) or assessment only (n=81). Outcomes will be assessed immediately post-intervention and at 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age
* Binge drinking in a typical week
* Any form of alcohol-induced memory impairment in the past month at baseline

Exclusion Criteria:

* Psychiatric disorder requiring immediate clinical attention (e.g., psychosis, suicidal ideation with intent and plan)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 169 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Recruitment | Baseline
  % of screened participants who (yes/no) complete the baseline assessment (no specific tool)
Retention | 3-month follow-up
  % of randomized participants who (yes/no) complete 3-month follow-up assessment (no specific tool)
Acceptability | 1 month follow-up
  Measured using the 8-item Client Satisfaction Questionnaire. Scored from 1 to 4, with higher scores indicating greater satisfaction with treatment.
Frequency of high-intensity drinking | Change from baseline to follow-up (1 and 3 months)
  Measured using the Daily Drinking Questionnaire, which asks participants to indicate how many standard drinks they consumed on each day of a typical week in the past month.
Peak BAC | Change from baseline to follow-up (1 and 3 months)
  Measured using the Daily Drinking Questionnaire, which asks participants to indicate the maximum number of drinks consumed on one occasion in the past month.
Frequency of blackouts | Change from baseline to follow-up (1 and 3 months)
  Measured using the 8-item Alcohol-Induced Blackout Measure-2 (ABOM-2). Items are scored from 0 to 4, with higher scores indicating more frequent blackout experiences.
Alcohol-related consequences | Change from baseline to follow-up (1 and 3 months)
  Measured using the 24-item Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ). Items scores yes/no, with higher scores indicating a greater number of consequences in the past month.

SECONDARY OUTCOMES:
Sexual coercion | Difference in likelihood baseline vs 3 months
  % of people indicating they (a) were coerced into sexual activity or (b) coerced someone else into sexual activity in the past 3 months
Emergency department visits | Difference in likelihood baseline vs 3 months
  % of people indicating they visited the emergency department in the past 3 months
Blackout susceptibility | Change from baseline to follow-up (1 and 3 months)
  How likely is it that you will lose memory of drinking events as a result of alcohol use in the next 30 days? Scored on a Likert scale, with higher scores indicating more susceptibility.
Blackout severity | Change from baseline to follow-up (1 and 3 months)
  If I were to have a blackout, bad things would happen. Scored on a Likert scale, with higher scores indicating more negative attitudes.
Costs/benefits of drinking | Change from baseline to follow-up (1 and 3 months)
  Measured using the Cunningham et al. (1997) scale of 16 benefits and 16 costs of decreasing alcohol use. Responses range 1 (not important) to 5 (extremely important).
Blackout self-efficacy | Change from baseline to follow-up (1 and 3 months)
  % confidence that participants could avoid a blackout, if they wanted to do so
Sleep disturbance | Change from baseline to follow-up (1 and 3 months)
  Measured using the Insomnia Severity Index. Items scored 0 to 4, with higher scores indicating more severe insomnia.
Mood | Change from baseline to follow-up (1 and 3 months)
  Measured using the Positive and Negative Affect Schedule. Scores range 1 (very slightly or not at all) to 5 (extremely), with higher scores indicating more positive/negative mood.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Miller, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, individual-level data will be deposited online via the NIAAA Data Archive (NIAAADA). De-identified data, the survey protocol and instrument, and analysis code will also be made available to other qualified investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon study completion
Access Criteria: NOT-AA-19-020
URL: https://grants.nih.gov/grants/guide/notice-files/NOT-AA-19-020.html